CLINICAL TRIAL: NCT04019678
Title: Breast Carcinoma T1-T2-T3 / cN +: Axillary Conservation of Lymph Nodes in the Presence of Micro Metastases in Sentinel Lymph Node, in cN- After Neoadjuvant Chemotherapy - Studio NEONOD 2
Brief Title: Breast Cancer: Axillary Conservation After Neoadjuvant Chemotherapy in Micro Metastatic Sentinel Lymph Nodes.
Acronym: NEONOD2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 651
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: experimental (Experimental): patients with micro metastatic sentinel lymph node and/or parasentinella lymph node (ypN1mi). Axillary dissection is not performed.
  Interventions: Procedure: Omission of Axillary dissection
- Group 2: standard (Active Comparator): patients with negative sentinel lymph node (ypN0) or with ITC finding (ypN0 / YpN0 (i +)). Axillary dissection is not performed as standard treatment.
  Interventions: Procedure: Omission of Axillary dissection

INTERVENTIONS:
Procedure: Omission of Axillary dissection — In Group 1 and 2: Axillary dissection won't be performed

SUMMARY:
Italian multicentric non inferiority clinical study to verify whether the omission of axillary lymph node intervention in patients with SLN (Sentinel Lymph Nodes) ypN1mi after NAC (Neo Adiuvant Chemotherapy) does not lead to a significant deterioration in survival or in the risk of regional or distant recurrence, compared to patients with negative SLN (SLN ypN0) after NAC ,where the omission of axillary treatment is currently the standard treatment.

DETAILED DESCRIPTION:
The study includes patients with cN+ positive axillary lymph nodes at initial diagnosis and who also have negative clinical and instrumental evaluation after NAC. Based on the sentinel lymph nodes definitive histological evaluation patients are allocated in one of the 2 comparison groups (Group 1 experimental or Group 2 standard) or in Group 3 internal control group. Group 3 is not used in statistical comparison with the other two groups but it's aim is to evaluate the appropriateness of the cases.

Referring to bio-pathologic characteristics after surgery patients will receive:

* no further treatment
* complementary radiotherapy
* adjuvant medical therapy (hormonal therapy and/or biological therapy)

Irradiation:

Group 1 (experimental) and Group 2 (standard): irradiation won't be performed neither in the axillary region nor in the other lymph node stations

Group 3 (internal control): after conservative or radical surgery, patients will be subjected to loco-regional irradiation according to Guidelines.

Duration:

Patients enrollment in the study protocol will last for 3 years. Patients will have to be followed for the subsequent 5 years during which they will have to undergo to periodic visits and follow-up checks provided for by the current standard guidelines:

* clinical examination every six months for the first 5 years
* mammography and breast ultrasound yearly
* axillary ultrasound yearly

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ≤75 years
2. Breast carcinoma with infiltrating histotype
3. Tumor size: cT1 - cT2 - cT3
4. Positive axillary lymph nodes (cN +) at the initial diagnosis by clinical, ultrasound and cyto-microhistology evaluation
5. Neoadjuvant chemotherapy performed
6. Negative axillary lymph nodes (cN-) from the NAC by clinical and ultrasound assessment
7. Absence of distant metastases (M0)
8. Negative medical history for previous infiltrating breast cancer

Exclusion Criteria:

1. Current pregnancy or lactation status
2. Inflammatory breast cancer
3. In situ breast cancer
4. Synchronous contralateral breast cancer
5. Co-morbidity and/or medical disorder precluding any adjuvant therapy
6. Co-morbidity and/or medical/mental disorder making impossible making a regular follow-up
7. Other cancers in the previous 3 years (except forcarcinoma in situ of the uterine cervix, basalioma, squamous cell carcinoma or non-melanoma skin cancer)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2027-06-21 (Estimated); Study Completion 2027-06-21 (Estimated)

PRIMARY OUTCOMES:
Disease-free or death-free survival for any reason (DFS) | 5 years of follow up after surgery
  Evaluating whether in patients operated for breast cancer (cT1-T2-T3) with sentinel node micrometastases (SLNypN1mi) after neoadjuvant chemotherapy (NAC), the preservation of axillary lymph nodes is not associated with a clinically relevant prognostic deterioration using Kaplan-Meier Product Limit Estimator and the log-rank test

SECONDARY OUTCOMES:
Global Survival (OS) | 5 years of follow up after surgery
  Kaplan-Meier Product Limit Estimator and the log-rank test
Regional Disease Free Survival (RDFS) | 5 years of follow up after surgery
  Kaplan-Meier Product Limit Estimator and the log-rank test
Disease-free distance survival (DDFS) | 5 years of follow up after surgery
  Kaplan-Meier Product Limit Estimator and the log-rank test

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tinterri, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy